CLINICAL TRIAL: NCT03954951
Title: Approaches to Reduce Clinical Inertia in Hypertension Management in Primary Care in the Dominican Republic
Brief Title: Approaches to Reduce Clinical Inertia in Hypertension in the Dominican Republic
Acronym: ARCH DR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit/maintain participants for intervention
Sponsor: Yale University (Other)
Collaborators: Instituto Tecnológico de Santo Domingo (INTEC) (Other)
Responsible Party: Principal Investigator, Robert McNamara, Associate Professor of Medicine (Cardiology), Yale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000023037
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Hypertension
Keywords: hypertension; blood pressure; clinical inertia; randomized clinical trial; uncontrolled hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel-group, cluster randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The clinicians in the control group will continue usual care without intervention. They will not receive the online course or performance feedback reports.
- Intervention group (Active Comparator): The primary care physicians will receive access to an online course on hypertension management based on the ACC/AHA and ESC guidelines. They will also receive feedback reports on their performance on hypertension management for 16 weeks.
  Interventions: Other: Multimodality behavioral strategy

INTERVENTIONS:
Other: Multimodality behavioral strategy — * On-line course on hypertension management based on the new ACC/AHA and ESC/ESH guidelines on hypertension management.
  * Weekly performance feedback reports: will include percent of patients with uncontrolled hypertension and among this group percent of visits where no change in medication was made. It will also include a comparative assessment of the performance of the physicians compared with their colleagues in the province.
  Arms: Intervention group

SUMMARY:
The purpose of this cluster randomized control trial is to test whether a multimodality strategy that includes an educational on-line course and performance feedback reports is effective to reduce clinical inertia in the management of hypertension in rural primary care clinics in the Dominican Republic.

DETAILED DESCRIPTION:
Proper control of elevated blood pressure (BP) is complex due to the large number of factors associated with therapy such as patient lifestyle, therapeutic adherence and access to health care, especially in low and middle income countries. More recently another obstacle has been described; clinical inertia, defined as the failure of clinicians to initiate or intensify antihypertensive therapy despite elevated BP levels not at goal. Suboptimal therapy is the most clinically important modifiable factor known to be associated with poor BP control. Reducing clinical inertia is of significant relevance, since a proper control of hypertension can reduce mortality from coronary heart disease and mortality from cerebrovascular disease.

Our hypothesis is that a multimodality strategy that includes an on-line course on updated guidelines on hypertension management and feedback performance reports is effective to reduce clinical inertia in the management of hypertension in rural primary care clinics in the Dominican Republic.

To test this hypothesis, this study will enroll eight clinics in rural neighborhoods of the Peravia province. These are government-funded small clinics that provide primary care and preventive services and are staffed with 2-3 primary care physicians. Eight clinics will be randomized at a 1:1 ratio into a control group and and intervention group. We anticipate over 500 patients from these clinics will be included.

The primary care physicians in the intervention group will be provided with an on-line course and weekly performance feedback reports, based on the new American College of Cardiology/American Heart Association (ACC/AHA) and European Society of Cardiology/European Society of Hypertension (ESC/ESH) hypertension guidelines. The performance feedback reports will include percent of patients with uncontrolled hypertension and among this group percent of visits where intensification in anti-hypertensive therapy was made. It will also include a comparative assessment of the performance of the physicians compared to their colleagues. The control group will continue to follow the current usual care without intervention. The total intervention and follow-up time will be 16 weeks.

ELIGIBILITY:
Inclusion Criteria for Clinics:

* Primary care clinics in rural areas of the Peravia province with primary care physicians (general practitioners, family medicine, internists).

Inclusion Criteria for Patients:

* Adult patients over age 18 who receive primary care at the participating clinics with history of hypertension or with blood pressure >130/80 mmHg during the visit

Exclusion Criteria for patients:

* Pregnant patients
* Patients under age 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Proportion of visits with clinical inertia | 16 weeks
  Clinical inertia will be designated to visits where BP was uncontrolled (BP ≥140/90 or ≥130/80 in patients with comorbidities) where no intensification of therapy was done or no justification for deferring intensification was documented.

SECONDARY OUTCOMES:
Percentage of patients on guideline concordant hypertension management | 16 weeks
  When clinical action was taken during the visit, the appropriateness of the therapy will be evaluated according to the most recent AHA/ACC and ESC/ESH hypertension recommendations. Initial choice of antihypertensive drug therapy will be deemed appropriate if it is a thiazide diuretic, calcium channel blocker, angiotensin-converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB).
Percentage of clinic visits with controlled blood pressure | 16 weeks
  The percentage of patients with controlled blood pressure (<140/90 and <130/80 with comorbidities) will be compared between intervention and control group/
Percentage of clinic visits where counseling on lifestyle modifications was provided | 16 weeks
  Lifestyle modification counseling include: changes on diet, decrease salt intake, physical activity, alcohol intake and smoking cessation.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Tecnologico de Santo Domingo, Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: No